CLINICAL TRIAL: NCT06833177
Title: Eighteen Months Clinical Evaluation of Hybrid Ceramic Inlays Cemented with Giomer Based Self-adhesive Resin Cement Versus Resin-based Cement in Carious Posterior Teeth: Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Ceramage Inlays Cemented with Beautilink Self-Adhesive Resin Cement Versus Rely X Resin Cement in Carious Posterior Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Ahmed Gomaa, MSc. 2024, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20091993
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Caries Class Ii
Keywords: Inlays; Ceramage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cementation via Beautilink SA cement (Experimental): Ceramage inlays will be cemented using Beautilink SA cement
  * To enhance the adhesion, adhesive bonding agent BeautiBond Xtreme, Shofu will be applied on the tooth and cured according to the manufacturer's instructions.
  * Press the plunger of the auto-mix syringe of Beautilink SA to dispence the cement on the adhesive surface of the restoration.
  * Using a light-curing unit to cure each surface and marginal areas for 10 seconds. For areas where the light cannot reach, or when using opaque cement, hold the restoration in place for approximately 5 minutes after light-curing to allow for chemical curing.
  Interventions: Other: Beautilink SA cement
- Cementation via RelyX resin cement (Active Comparator): Ceramage inlays will be cemented using RelyX resin cement
  * To enhance the adhesion, adhesive bonding agent 3M™ Scotchbond™ Universal Plus Adhesive will be applied on the tooth and cured according to the manufacturer's instructions.
  * Application of 3M™RelyX™ Universal Resin Cement into the cavity
  * Using a light-curing unit to cure each surface and marginal areas for 10 seconds. For areas where the light cannot reach, or when using opaque cement, hold the restoration in place for approximately 6 minutes after light-curing to allow for chemical curing.
  Interventions: Other: RelyX resin cement

INTERVENTIONS:
Other: Beautilink SA cement — According to the manufacturer's instructions (BeautiLink SA - Shofu USA)
  * To enhance the adhesion, adhesive bonding agent BeautiBond Xtreme, Shofu will be applied on the tooth and cured according to the manufacturer's instructions.
  * Press the plunger of the auto-mix syringe of Beautilink SA to dispence the cement on the adhesive surface of the restoration.
  * Seat the restoration in the cavity and apply proper pressure after using Teflon to protect the adjacent teeth and help in the removal of the excess material.
  * Light-cure the excess material for 1-2 sec with a light-curing unit followed by removal of the tack-cured material with a probe.
  * Using a light-curing unit to cure each surface and marginal areas for 10 seconds. For areas where the light cannot reach, or when using opaque cement, hold the restoration in place for approximately 5 minutes after light-curing to allow for chemical curing.
  Arms: Cementation via Beautilink SA cement
Other: RelyX resin cement — According to the manufacturer's instructions (Espe).
  * To enhance the adhesion, adhesive bonding agent 3M™ Scotchbond™ Universal Plus Adhesive will be applied on the tooth and cured according to the manufacturer's instructions.
  * Application of 3M™RelyX™ Universal Resin Cement into the cavity
  * Seat the restoration in the cavity and apply proper pressure after using Teflon to protect the adjacent teeth and help in the removal of the excess material.
  * Light-cure the excess material for 2-3 sec with a light-curing unit followed by removal of the tack-cured material with a probe.
  * Using a light-curing unit to cure each surface and marginal areas for 10 seconds. For areas where the light cannot reach, or when using opaque cement, hold the restoration in place for approximately 6 minutes after light-curing to allow for chemical curing.
  Arms: Cementation via RelyX resin cement

SUMMARY:
Minimally invasive bonded partial restorations have become a crucial component of contemporary dental treatments. They address the shortcomings of direct restorations and provide patients with a less damaging alternative to full coverage restorations, which can be more harmful to the dental structure. Indirect inlay composite restorations have become a popular choice in restorative dentistry due to their aesthetic appeal and durability. These restorations allow for the preservation of tooth structure while utilizing the mechanical advantages of modern adhesive technology, which can reinforce the weakened compromised tooth structure.

The use of different adhesive materials with Ceramage can significantly influence the success of the restoration. Adhesive materials play a crucial role in ensuring a strong bond between the indirect restoration and the tooth structure. Additionally, the choice of adhesive material can also affect the ease of the cementation process. Self-adhesive resin cement simplifies the procedure by eliminating the need for separate bonding agents, thus reducing the risk of technique sensitivity which can lead to more consistent clinical outcomes and improved patient satisfaction.

Overall, the combination of Ceramage with appropriate adhesive materials offers a reliable and aesthetically pleasing solution for indirect inlay composite restorations, enhancing both the biological, functional and esthetic outcomes of dental treatments.

ELIGIBILITY:
Inclusion Criteria:

* Posterior vital tooth with a large carious lesion (ICDAS 4/5)
* Posterior vital tooth with a broken restoration that should be replaced (ICDAS 4-7/5-7).
* Vital, periodontally sound and with positive reaction to cold stimulus.
* Fully erupted posterior molar in normal functional occlusion with natural antagonist and adjacent teeth.

Exclusion Criteria:

* Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
* Non-vital teeth, Fractured or cracked teeth.
* Endodontically treated teeth.
* Periodontally affected teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance assessing Biological, Mechanical and Esthetic Parameters Using Modified USPHS Criteria | T0: 12 months T1: 18 months
  Alpha being the best results and Charlie being the worst results

IPD SHARING:
Plan to Share IPD: Undecided